CLINICAL TRIAL: NCT04227119
Title: Hemodynamics Measurement in Radiofrequency Catheter Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Anand D Shah, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00116832
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Arrhythmia
Keywords: Cardiology; Electrophysiology
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Irrigated ablation catheter and 5F balloon tipped PA catheter (Experimental): Participants undergoing cardiac ablation will have cardiac pressures measured with an irrigated ablation catheter (standard protocol for this procedure) and a 5F balloon tipped pulmonary artery (PA) catheter (for study purposes only).
  Interventions: Device: Irrigated ablation catheter; Device: Balloon tipped PA catheter

INTERVENTIONS:
Device: Irrigated ablation catheter — After completion of ablation, the ablation catheter will be serially positioned in the cardiac chambers (either the left or right side of the heart). The stop cock will be turned to the pressure transducer and waveforms will be stored corresponding to each chamber.
Device: Balloon tipped PA catheter — After removal of the irrigated ablation catheter, a 5F balloon tipped PA catheter which will be positioned under fluoroscopic guidance in each previously evaluated chamber and the chambers will be measured again.

SUMMARY:
This study will occur in patients undergoing routine cardiac ablation of his/her arrhythmia with planned use of an irrigated ablation catheter. The main objective of this study is to take intracardiac pressure measurements and pressure waveforms with both a "gold standard" balloon tipped pulmonary artery catheter placed for this study and an irrigated ablation catheter placed as standard of care for the procedure.

DETAILED DESCRIPTION:
Measuring internal heart pressures allows for the assessment and diagnosis of a variety of cardiac conditions which are commonly found in patients undergoing catheter ablation, including congestive heart failure, diastolic dysfunction, and valvular heart disease. Currently it is unknown if taking pressure measurements with the ablation catheter is accurate and it is not standard practice to insert the additional 'gold standard' pressure sensing catheter. Catheter ablation of cardiac arrhythmia is performed to offer symptomatic relief from a variety of atrial, ventricular and atrio-ventricular rhythms. Irrigated ablation catheters are commonly used for ablation of arrhythmias arising from the left heart and coronary sinus. These catheters contain internal channels allowing for infusion of an external fluid directly to the tip of the catheter, where the fluid is sprayed through numerous end holes allowing for cooling of the catheter ablation tip.

Fluid filled catheters are also the primary tool utilized to assess intravascular and intracardiac pressures and hemodynamics in the cardiac catheterization suite and intensive care unit. However, the fluid filled catheters commonly used for these assessments are single lumen with a single end hole and generally have a larger minimal diameters compared to the ablation catheter. "Dampening" of pressure waveforms are observed in smaller diameter catheters and may lead to underestimation of peak pressure and overestimation of the nadir pressure gradient. It is unknown if transduction of pressures from the tip of an irrigated ablation catheter will yield equivalent results compared to use of a single 5 French (5F) sized lumen catheter.

This study will seek to enroll patients already scheduled to have a cardiac ablation for a clinical arrhythmia at Emory University Hospital. After completion of the standard ablation, the ablation catheter will be positioned in the heart and pressures will be measured. Next, a standard pressure sensing catheter will be positioned in the same area in the heart and pressures will be measured. The pressure values for each heart chamber assessed will be compared between the catheters. The purpose of this study is to test the hypothesis that transduction of intracardiac pressures using an irrigated ablation catheter placed as standard of care for the ablation procedure is equivalent to transduction of pressures using a standard 5F balloon tipped PA catheter placed only for this research study.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing routine cardiac ablation of his/her arrhythmia with planned use of an irrigated ablation catheter

Exclusion Criteria:

* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand D Shah, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the patient population at Emory University Hospital and the Emory Clinic, in Atlanta, Georgia who were scheduled to have a routine cardiac ablation using an irrigated ablation catheter for treatment of arrhythmia. Participants were enrolled between January 23, 2020 and May 18, 2020.
Groups:
- Irrigated Ablation Catheter and Balloon Tipped PA Catheter: Participants undergoing cardiac ablation had cardiac pressures measured with an irrigated ablation catheter (standard protocol for this procedure) and a 5 French (5F) sized balloon tipped pulmonary artery (PA) catheter (for study purposes only).
  The catheter will be positioned in either the left or right side of the heart.
Period: Overall Study
Arm/Group | Irrigated Ablation Catheter and Balloon Tipped PA Catheter
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Irrigated Ablation Catheter and Balloon Tipped PA Catheter: Participants undergoing cardiac ablation had cardiac pressures measured with an irrigated ablation catheter (standard protocol for this procedure) and a 5F balloon tipped pulmonary artery (PA) catheter (for study purposes only).
Arm/Group | Irrigated Ablation Catheter and Balloon Tipped PA Catheter
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Indication for Ablation [Count of Participants; unit: Participants]
  Atrial fibrillation | 9
  Ventricular tachycardia | 2
Ejection Fraction [Mean (Standard Deviation); unit: percentage of blood pumped] | 47.3 (16.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (4.6)
Type of Atrial Fibrillation [Count of Participants; unit: Participants]
  Paroxysmal atrial fibrillation | 4
  Persistent atrial fibrillation | 5
  No atrial fibrillation | 2

OUTCOME MEASURES:

1. Primary Outcome: Systolic Pressure Value
Description: The systolic pressure values for atrium and ventricle heart chambers are presented for the irrigated ablation catheter derived measurements and the balloon tipped PA catheter measurements.
Time Frame: Day 1 (during procedure)
Population: Participants had the ablation catheter positioned in only one side of the heart. Nine participants had measurements obtained from the left atrium and ventricle chambers, and two participants had measurements obtained from the right atrium and ventricle chambers.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Irrigated Ablation Catheter: Participants undergoing cardiac ablation had cardiac pressures measured with an irrigated ablation catheter (standard protocol for this procedure).
- Balloon Tipped PA Catheter: Participants undergoing cardiac ablation had cardiac pressures measured with a 5F balloon tipped pulmonary artery (PA) catheter (for study purposes only).
Arm/Group | Irrigated Ablation Catheter | Balloon Tipped PA Catheter
Number analyzed (Participants) | 11 | 11
millimeters of mercury (mmHg)
  Left atrium: number analyzed (Participants) | 9 | 9
  Left atrium | 26.5 (6.4) | 27.75 (7.4)
  Right atrium: number analyzed (Participants) | 2 | 2
  Right atrium | 16.6 (5.1) | 13.6 (6.3)
  Left ventricle: number analyzed (Participants) | 9 | 9
  Left ventricle | 114.6 (33.4) | 105.9 (30.4)
  Right ventricle: number analyzed (Participants) | 2 | 2
  Right ventricle | 42.8 (3.6) | 54.1 (2.8)

2. Primary Outcome: Diastolic Pressure Value
Description: The diastolic pressure values for ventricle heart chambers are presented for the irrigated ablation catheter derived measurements and the balloon tipped PA catheter measurements.
Time Frame: Day 1 (during procedure)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Irrigated Ablation Catheter | Balloon Tipped PA Catheter
Number analyzed (Participants) | 11 | 11
mmHg
  Left ventricle: number analyzed (Participants) | 9 | 9
  Left ventricle | 15.3 (4.0) | 17.3 (3.2)
  Right ventricle: number analyzed (Participants) | 2 | 2
  Right ventricle | 20.2 (5.2) | 15.8 (4.6)

3. Post Hoc Outcome: Systolic Pressure Per Millisecond
Description: The systolic pressure values per time, in milliseconds (ms), for the left ventricle chamber is presented for the irrigated ablation catheter derived measurements and the balloon tipped PA catheter measurements.
Time Frame: Day 1 (during procedure)
Population: This analysis includes the nine participants had measurements obtained from the left ventricle chamber.
Measure: Mean (Standard Deviation); unit: mmHg/ms
Arm/Group | Irrigated Ablation Catheter | Balloon Tipped PA Catheter
Number analyzed (Participants) | 9 | 9
mmHg/ms | 0.49 (0.15) | 0.53 (0.11)

ADVERSE EVENTS:
Time Frame: Data on adverse events will be collected from the start of the procedure through the end of the procedure on Day 1 of the study.
Arm/Group | Irrigated Ablation Catheter | Balloon Tipped PA Catheter
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04227119/Prot_SAP_000.pdf